CLINICAL TRIAL: NCT00564967
Title: A Comparison Between Internet-based Self-help Therapy and Group Therapy for Social Phobia - A Clinical Equivalence Trial Using Cognitive Behavioural Therapy (CBT)
Brief Title: A Comparison Between Internet Therapy and Group Therapy for Social Phobia - A Trial Using Cognitive Behavioural Therapy
Acronym: IS1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Nils Lindefors, MD, PHD, professor, Stockholm County Council and Karolinska Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IS1; Dnr 2005/178-31
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2009-08

CONDITIONS: Social Phobia
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CBT via the Internet
  Interventions: Behavioral: CBT via the Internet
- 2 (Experimental): 15 weeks, CBT group therapy, 1 session/week (2.5 hours).
  Interventions: Behavioral: CBT group therapy

INTERVENTIONS:
Behavioral: CBT via the Internet — 15 weeks, patients learn about CBT primarily thru a self-help book published on teh Internet, Minimal therapy contact via e-mail(10 minutes/week),
  Arms: 1
Behavioral: CBT group therapy — 15 weeks, 1 session/week, (2,5 hours.)
  Arms: 2

SUMMARY:
Social phobia is one of the most prevalent anxiety disorders in the western world. Cognitive behavioural therapy (CBT) is the psychological treatment that has the largest empirical support. However, the availability to CBT is very limited in Sweden due to lack of therapists with proper training. Therefore it is important to evaluate alternative forms of treatment that are more time efficient. One of these methods is Internet based self-help therapy, which has proven to be an effective treatment for social phobia.

To the investigator´s knowledge, no study has yet directly compared live-CBT to Internet therapy. The aim of the present study is to compare the effect of live CBT vs CBT delivered via the Internet. The study is considered to be an equivalence trial. 128 patients will be randomly assigned to one of the two treatment conditions. The primary outcome measure is Liebowitz Social Anxiety Scale (LSAS).

ELIGIBILITY:
Inclusion Criteria:

* Must have a primary diagnosis of social phobia

Exclusion Criteria:

* Substance abuse during the last 6 months
* Other dominating diagnosis (not phobic personality disorder)
* A history of bipolar disorder or psychosis
* Major depression according to DSM-IV and >20 on madrs-s
* Risk of suicide
* Start of medication or change of dosis during the last 2 months
* Other parallel psychological treatment
* Previous CBT (last 3 years) for social phobia

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS)

SECONDARY OUTCOMES:
SIAS, SPS,QOLI,MADRS-S, BAI,ASI,CGI, WQ, GAF, TIC-P, SSP

CONTACTS AND LOCATIONS:
Overall Officials: nils lindefors, Principal Investigator — Karolinska Institutet
Locations (1):
- Psykiatri Sydväst, Stockholm County Council, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Andersson E, Ruck C, Lavebratt C, Hedman E, Schalling M, Lindefors N, Eriksson E, Carlbring P, Andersson G, Furmark T. Genetic polymorphisms in monoamine systems and outcome of cognitive behavior therapy for social anxiety disorder. PLoS One. 2013 Nov 15;8(11):e79015. doi: 10.1371/journal.pone.0079015. eCollection 2013. PMID 24260145
- [Derived] Hedman E, Andersson E, Ljotsson B, Andersson G, Andersson E, Schalling M, Lindefors N, Ruck C. Clinical and genetic outcome determinants of Internet- and group-based cognitive behavior therapy for social anxiety disorder. Acta Psychiatr Scand. 2012 Aug;126(2):126-36. doi: 10.1111/j.1600-0447.2012.01834.x. Epub 2012 Feb 9. PMID 22320999
- [Derived] Hedman E, Andersson G, Ljotsson B, Andersson E, Ruck C, Mortberg E, Lindefors N. Internet-based cognitive behavior therapy vs. cognitive behavioral group therapy for social anxiety disorder: a randomized controlled non-inferiority trial. PLoS One. 2011 Mar 25;6(3):e18001. doi: 10.1371/journal.pone.0018001. PMID 21483704
- See also: Information about the study and how to enroll is provided — http://www.internetpsykiatri.se